CLINICAL TRIAL: NCT03291639
Title: Functional Plasticity of Human IL-17-producing CD8+ T Cells
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH106-REC3-107
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: IL-17+ CD8 T Cells in Cancer Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human Tc17 cells (IL-17-producing CD8+ T cells) have been found to contribute to different kinds of human inflammatory and malignant diseases. Previous studies indicate that Tc17 cells can convert to Tc1 cells (IFN-γ-producing CD8+ T cells) in tumor bearing mice to exert anti-tumor effect. Base on these results in murine models, human Tc17 may have potential in developing cancer immunotherapy. However, there is limited evidence to reveal the characteristics and functional plasticity of human Tc17 cells. In this proposal, we aim to optimize the differentiation of Tc17 cells and then investigate whether the reprograming of Tc17 to Tc1 cells can promote the anti-tumor cytotoxicity. Preliminarily, we isolated CD8+ T cells from the peripheral blood mononuclear cells of healthy donors to induce Tc17 differentiation. Human CD8+ T cells were stimulated with anti-CD3/anti-CD28 antibodies, TGF-β, IL-1β, IL-6, IL-23, IL-2, anti-IFN-γ, and anti-IL-4 antibodies. After 10 days in culture, there were 4% of IL-17A+IFN-γ- and 7% of IL-17A+IFN-γ+ CD8+ T cells. However, IFN-γ+ CD8+ T cells still represented high percentage, although it's significantly lower than that in Tc1 cells. Our preliminary study demonstrated that Tc17 cells expressed lower levels of cytotoxic molecules than Tc1 cells. We will further test if the expressions of cytotoxic molecules, including perforin and granzyme B, and EOMES will be enhanced by various cytokines. Ultimately, we will evaluate the functional plasticity of Tc17 cells under various cytokine stimulation. Collectively, success of this project will establish more insight for human Tc17 cells and provide the information for future developing human CD8+ T cell-mediate immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients

Exclusion Criteria:

* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy donors and 20 cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Functional plasticity of IL-17+ CD8 T cells | culture cells for 16 days
  To skew human IL-17+ CD8 T cells and add specific cytokines to convert IL-17 CD8 T cells to IFN-gamma CD8 T cells

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan